CLINICAL TRIAL: NCT03459092
Title: A Pragmatic, Randomized, Non-inferiority Trial Comparing the Effectiveness of Botulinum Toxin-based Treatment With Conventional Strabismus Surgery in Acquired Esotropia.
Brief Title: Botox Instead of Strabismus Surgery (BISS)
Acronym: BISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33IC30 173533
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acquired Esotropia
Keywords: Botulinum toxin, strabismus surgery, binocular vision
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botox-based treatment regimen (Experimental): First intervention is a Botulinum toxin type A injection. If further treatment is necessary, strabismus surgery can be performed.
  Interventions: Drug: Botulinum toxin type A; Procedure: Strabismus surgery
- Surgery-based treatment regimen (Active Comparator): First intervention is strabismus surgery. If further treatment is necessary, strabismus surgery can be repeated.
  Interventions: Procedure: Strabismus surgery

INTERVENTIONS:
Drug: Botulinum toxin type A — Botulinum toxin injection in the horizontal extraocular muscles.
  Arms: Botox-based treatment regimen
Procedure: Strabismus surgery — Strabismus surgery on the horizontal extraocular muscles

SUMMARY:
The purpose of the study is to evaluate if strabismus can be successfully treated requiring less surgical interventions with a Botox-based treatment regimen compared to a purely surgery based treatment regimen.

Experimental arm: Botulinum toxin injection in the horizontal extraocular muscles.

Control (active comparator) arm: Strabismus surgery on the horizontal extraocular muscles. No investigational product is used.

In Switzerland the standard procedure for treating large angle esotropia is surgery, which is performed on the horizontal eye muscles that may be either recessed or shortened leading to reduced or increased muscle function respectively.

As an alternative to strabismus surgery, botulinum toxin (Botox) can be applied in extraocular muscles. Botox prevents the release of acetylcholine in the synaptic cleft and thereby blocks the neuromuscular transmission thus inducing a palsy.

Current evidence on the use of Botox in strabismus is incoherent, is poorly supported by basic research findings and leaves dedicated clinicians in the dark. The objective is to shed light into this field of clinical research, which may help to guide future pediatric ophthalmologists in their management of strabismic patients. In a best case scenario, the results from this trial will prevent strabismus operation for many children with acquired large angle esotropia.

DETAILED DESCRIPTION:
Patients with acquired large angle esotropia (an inward deviation of the ocular axis by more than 5°) that develops after one year of age have a potential to regain binocular vision if a retinal image appears on corresponding retinal areas of both eyes. The main goal of therapy in these patients is the restoration of binocular vision.

In Switzerland the standard procedure for treating large angle esotropia is surgery, which is performed on the horizontal eye muscles that may be either recessed or shortened leading to reduced or increased muscle function respectively.

As an alternative to strabismus surgery, botulinum toxin (Botox) can be applied in extraocular muscles. Botox prevents the release of acetylcholine in the synaptic cleft and thereby blocks the neuromuscular transmission thus inducing a palsy.

Current evidence on the use of Botox in strabismus is incoherent, is poorly supported by basic research findings and leaves dedicated clinicians in the dark. The goal is to shed light into this field of clinical research, which may help to guide future pediatric ophthalmologists in their management of strabismic patients.

The goal of the study is to test if, with a botulinum-toxin-based treatment regimen, strabismus can be successfully treated requiring less surgical interventions.

The primary objective is to test if the Botox-based treatment regimen is not inferior to surgical treatment in terms of orthotropic success. If this is shown, the number of surgeries required will be compared between the two groups (main secondary objective).

The hypothesis is that the Botox-based treatment regimen, which permits performance of rescue surgery, is successful in a similar proportion of patients as the purely surgical approach. The second hypothesis is that only about 20% of patients treated with Botox require surgery at all as compared to about 10% of patients in the surgical arm that need a second surgery.

Analysis of the primary outcome The proportion of orthotropic success for both groups will be calculated with a corresponding 95% confidence interval. For the comparison between the two groups, the stratified risk difference for the stratification factors used in randomization will be calculated with a corresponding one-sided lower 95% confidence limit. If the lower limit lies above -12%, non-inferiority will be claimed.

Analysis of the main secondary outcome The proportion of second interventions for both groups will be calculated with a corresponding 95% confidence interval. For the comparison between the two groups, a stratified risk difference for the stratification factors used in randomization will be calculated with a corresponding one-sided upper 95% confidence limit. If the upper limit lies below 40% and if non-inferiority for the primary outcome could be demonstrated, a clinical benefit of the new treatment will be claimed.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent of trial participant and/or legal representative documented per signature
2. Age > 1 year and <17 years
3. Esotropia > 10Prisms
4. Indication for an intervention (either Botox or surgery) has been made.
5. Any of the following:

   * Presence of a secondary strabismus from binocular disruption the cause of the binocular disruption is no longer present
   * Decompensated microstrabismus
   * Decompensated phoria
   * Acute acquired esotropia
6. Positive test of binocular function at any time point in the past, including any of the following

   * Titmus test
   * Bagolini striated glasses test
   * Lang-stereo-test with correct naming of at least one panel
   * Good ocular alignment after 6 months of age on at least 2 photographs

Exclusion Criteria:

1. Known hypersensitivity to botulinum toxin
2. Known neuromuscular disorder
3. Known present neurological disorder affecting the central nervous system Including paresis on cranial nerves number 3, 4 and 6
4. Any of the following:

   * nystagmus
   * dissociated vertical deviation
5. Vertical deviation in any gaze direction greater than 5°
6. Incomitance with more than 5° of difference between the left and right horizontal gaze direction
7. Previous strabismus surgery
8. Previous Botulinum toxin treatment on extraocular muscles
9. Presence of ophthalmic pathologies significantly preventing binocular functions.

   A significant alteration of binocular function is assumed if vision is smaller than 0.1 or the visual field has a horizontal diameter of less than 20°.
10. Pregnancy. A negative pregnancy test before randomization is required for all women of child-bearing potential.
11. Preterm children born before 36 weeks of gestation.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2018-08-16 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with presence of binocular vision | At 18 months
  Presence of binocular vision is a binary variable set to yes when either of the following criteria is fulfilled:
  1. No eye movement can be observed in the simultaneous prism covertest, performed according to the study specific SOP for full orthoptic workup, for both eyes measured at distance. This proves orthotropia and thus binocular vision can be assumed.
  2. An esotropia of less than 5° is observed in the covertest at distance AND at near. In addition at least one binocular test demonstrates binocular vision. This proves compensated microstrabismus with anomalous retinal correspondence.
  Binocular tests:
  1. Lang-Stereotest
  2. Butterfly- Stereotest
  3. Titmus test
  4. Bagolini striated glasses test
  5. TNO-Test
  6. Pencil-Test

SECONDARY OUTCOMES:
Number of patients with second intervention | At 12 months, at 18 months
  Rescue surgery in Botox-based treatment arm and second surgery in surgery arm
Number of patients with binocular vision | At 12 months
  Presence of binocular vision is a binary variable set to yes when either of the following criteria is fulfilled:
  1. No eye movement can be observed in the simultaneous prism covertest, performed according to the study specific SOP for full orthoptic workup, for both eyes measured at distance. This proves orthotropia and thus binocular vision can be assumed.
  2. An esotropia of less than 5° is observed in the covertest at distance AND at near. In addition at least one binocular test demonstrates binocular vision. This proves compensated microstrabismus with anomalous retinal correspondence.
  Binocular tests:
  1. Lang-Stereotest
  2. Butterfly- Stereotest
  3. Titmus test
  4. Bagolini striated glasses test
  5. TNO-Test
  6. Pencil-Test
Number of patients with incomitance | At 12 months, at 18 months
  Incomitance is here defined as the absolute difference of strabismus angle measured with the alternate prism cover test at 25° left gaze and the angle measured at 25° right gaze
Number of patients with treatment-specific presence of binocular vision | At 12 months, at 18 months
  For this outcome patients with a second intervention are defined as failures (no).
Number of surgeries per participant | At 12 months, at 18 months
Number of surgeries needed per successful outcome | At 12 months, at 18 months
  Successful outcome = binocular vision
Change in strabismus angle, measured in percent | At 12 months, at 18 months
  Measured as percentage of preoperative deviation from baseline. The strabismus angle measured with the alternate prism cover test, performed in primary position at distance is used. Change of deviation in percent of preoperative deviation is calculated as follows:
  100*(preoperative deviation - postoperative deviation) / preoperative deviation
Binocular function, measured in arc seconds | At 12 months, at 18 months
  When binocular vision is present, the binocular function is the best stereoscopic acuity, measured in arc seconds, achieved for any of the below mentioned tests.
  1. Lang-Stereotest
  2. Butterfly- Stereotest
  3. Titmus test
  4. Bagolini striated glasses test
  5. TNO-Test
  6. Pencil-Test

OTHER OUTCOMES:
Total duration of binocular vision (exploratory outcome) | At 12 months, at 18 months
  The duration is calculated as the sum of time periods between consecutive assessments with presence of binocular vision.
Incidence of short-term adverse events (safety outcome) | Within two weeks of intervention
  Adverse event groups that will be evaluated separately are:
  * Ptosis
  * Double vision
  * Subjective post-treatment discomfort/pain
  * New vertical strabismus >1°
  * Limitations of ocular motility
Incidence of ocular adverse events | Within 18 months
Incidence of serious adverse events related to the treatment | Within 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Abegg, Professor, Principal Investigator — Bern University Hospital
Locations (8):
- Institut Ophtalmologique Sourdille Atlantique, Saint-Herblain, France
- Switzerland (7):
  - Basel University Hopital, Basel
  - Bern University Hospital, Bern
  - Geneva University Hospital, HUG, Geneva
  - Lausanne Univeristy Hospital, CHUV, Lausanne
  - Luzerner Kantonsspital, Lucerne
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Yes
The de-identified study dataset will be made publicly available for secondary analyses by publishing the data on a data sharing platform such as Dryad or BORIS, the public online data repository from the University of Bern.
Supporting Information: Study Protocol, SAP
Time Frame: Once the primary analysis is published.

REFERENCES:
- [Background] Scott AB. Botulinum toxin injection into extraocular muscles as an alternative to strabismus surgery. Ophthalmology. 1980 Oct;87(10):1044-9. doi: 10.1016/s0161-6420(80)35127-0. PMID 7243198
- [Background] Tejedor J, Rodriguez JM. Early retreatment of infantile esotropia: comparison of reoperation and botulinum toxin. Br J Ophthalmol. 1999 Jul;83(7):783-7. doi: 10.1136/bjo.83.7.783. PMID 10381663
- [Background] Tejedor J, Rodriguez JM. Retreatment of children after surgery for acquired esotropia: reoperation versus botulinum injection. Br J Ophthalmol. 1998 Feb;82(2):110-4. doi: 10.1136/bjo.82.2.110. PMID 9613374
- [Background] Lee J, Harris S, Cohen J, Cooper K, MacEwen C, Jones S. Results of a prospective randomized trial of botulinum toxin therapy in acute unilateral sixth nerve palsy. J Pediatr Ophthalmol Strabismus. 1994 Sep-Oct;31(5):283-6. doi: 10.3928/0191-3913-19940901-03. PMID 7837013
- [Background] Carruthers JD, Kennedy RA, Bagaric D. Botulinum vs adjustable suture surgery in the treatment of horizontal misalignment in adult patients lacking fusion. Arch Ophthalmol. 1990 Oct;108(10):1432-5. doi: 10.1001/archopht.1990.01070120080033. PMID 2222277
- [Background] de Alba Campomanes AG, Binenbaum G, Campomanes Eguiarte G. Comparison of botulinum toxin with surgery as primary treatment for infantile esotropia. J AAPOS. 2010 Apr;14(2):111-6. doi: 10.1016/j.jaapos.2009.12.162. PMID 20451851
- [Background] McNeer KW, Tucker MG, Spencer RF. Botulinum toxin management of essential infantile esotropia in children. Arch Ophthalmol. 1997 Nov;115(11):1411-8. doi: 10.1001/archopht.1997.01100160581010. PMID 9366672
- [Background] Lueder GT, Galli M, Tychsen L, Yildirim C, Pegado V. Long-term results of botulinum toxin-augmented medial rectus recessions for large-angle infantile esotropia. Am J Ophthalmol. 2012 Mar;153(3):560-3. doi: 10.1016/j.ajo.2011.08.019. Epub 2011 Oct 13. PMID 21996305
- [Background] Gursoy H, Basmak H, Sahin A, Yildirim N, Aydin Y, Colak E. Long-term follow-up of bilateral botulinum toxin injections versus bilateral recessions of the medial rectus muscles for treatment of infantile esotropia. J AAPOS. 2012 Jun;16(3):269-73. doi: 10.1016/j.jaapos.2012.01.010. PMID 22681945
- [Background] Baggesen K, Arnljot HM. Treatment of congenital esotropia with botulinum toxin type A. Acta Ophthalmol. 2011 Aug;89(5):484-8. doi: 10.1111/j.1755-3768.2009.01737.x. Epub 2009 Oct 30. PMID 19878118
- [Background] Campos EC, Schiavi C, Bellusci C. Critical age of botulinum toxin treatment in essential infantile esotropia. J Pediatr Ophthalmol Strabismus. 2000 Nov-Dec;37(6):328-32; quiz 354-5. doi: 10.3928/0191-3913-20001101-05. PMID 11392405
- [Background] Biglan AW, Burnstine RA, Rogers GL, Saunders RA. Management of strabismus with botulinum A toxin. Ophthalmology. 1989 Jul;96(7):935-43. doi: 10.1016/s0161-6420(89)32776-x. PMID 2771360
- [Background] Kushner BJ, Morton GV. A randomized comparison of surgical procedures for infantile esotropia. Am J Ophthalmol. 1984 Jul 15;98(1):50-61. doi: 10.1016/0002-9394(84)90188-0. PMID 6377903
- [Background] Helveston EM, Ellis FD, Schott J, Mitchelson J, Weber JC, Taube S, Miller K. Surgical treatment of congenital esotropia. Am J Ophthalmol. 1983 Aug;96(2):218-28. doi: 10.1016/s0002-9394(14)77790-6. PMID 6881245
- [Background] Scheiman M, Ciner E, Gallaway M. Surgical success rates in infantile esotropia. J Am Optom Assoc. 1989 Jan;60(1):22-31. PMID 2644332
- [Background] Hatt SR, Leske DA, Liebermann L, Holmes JM. Comparing outcome criteria performance in adult strabismus surgery. Ophthalmology. 2012 Sep;119(9):1930-6. doi: 10.1016/j.ophtha.2012.02.035. Epub 2012 Apr 26. PMID 22541935
- [Background] Wan MJ, Mantagos IS, Shah AS, Kazlas M, Hunter DG. Comparison of Botulinum Toxin With Surgery for the Treatment of Acute-Onset Comitant Esotropia in Children. Am J Ophthalmol. 2017 Apr;176:33-39. doi: 10.1016/j.ajo.2016.12.024. Epub 2017 Jan 3. PMID 28057455
- [Background] Dysli M, Keller F, Abegg M. Acute onset incomitant image disparity modifies saccadic and vergence eye movements. J Vis. 2015 Mar 18;15(3):12. doi: 10.1167/15.3.12. PMID 25788706
- [Background] Dysli M, Abegg M. Gaze-dependent phoria and vergence adaptation. J Vis. 2016;16(3):2. doi: 10.1167/16.3.2. PMID 26830708
- [Background] Mahan M, Engel JM. The resurgence of botulinum toxin injection for strabismus in children. Curr Opin Ophthalmol. 2017 Sep;28(5):460-464. doi: 10.1097/ICU.0000000000000408. PMID 28650877
- [Background] Pediatric Eye Disease Investigator Group; Christiansen SP, Chandler DL, Lee KA, Superstein R, de Alba Campomanes A, Bothun ED, Morin J, Wallace DK, Kraker RT. Tonic pupil after botulinum toxin-A injection for treatment of esotropia in children. J AAPOS. 2016 Feb;20(1):78-81. doi: 10.1016/j.jaapos.2015.09.011. PMID 26917081
- [Background] Pehere N, Jalali S, Mathai A, Naik M, Ramesh K. Inadvertent intraocular injection of botulinum toxin A. J Pediatr Ophthalmol Strabismus. 2011 Jan 25;48 Online:e1-3. doi: 10.3928/01913913-20110118-06. PMID 21261223
- [Background] Liu M, Lee HC, Hertle RW, Ho AC. Retinal detachment from inadvertent intraocular injection of botulinum toxin A. Am J Ophthalmol. 2004 Jan;137(1):201-2. doi: 10.1016/s0002-9394(03)00837-7. PMID 14700677
- [Background] Bradbury JA, Taylor RH. Severe complications of strabismus surgery. J AAPOS. 2013 Feb;17(1):59-63. doi: 10.1016/j.jaapos.2012.10.016. Epub 2013 Jan 23. PMID 23352718
- [Background] Ares C, Superstein R. Retrobulbar hemorrhage following strabismus surgery. J AAPOS. 2006 Dec;10(6):594-5. doi: 10.1016/j.jaapos.2006.04.005. Epub 2006 Oct 2. PMID 17189162
- [Background] Rowe FJ, Noonan CP. Botulinum toxin for the treatment of strabismus. Cochrane Database Syst Rev. 2017 Mar 2;3(3):CD006499. doi: 10.1002/14651858.CD006499.pub4. PMID 28253424
- [Background] Lyons CJ, Tiffin PA, Oystreck D. Acute acquired comitant esotropia: a prospective study. Eye (Lond). 1999 Oct;13 ( Pt 5):617-20. doi: 10.1038/eye.1999.169. PMID 10696312
- [Background] BURIAN HM, MILLER JE. Comitant convergent strabismus with acute onset. Am J Ophthalmol. 1958 Apr;45(4 Pt 2):55-64. doi: 10.1016/0002-9394(58)90223-x. No abstract available. PMID 13520873